CLINICAL TRIAL: NCT01833975
Title: Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Spinal Cord Injury . It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Spinal Cord Injury
Acronym: SCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, C0- Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00103
Record Dates: First submitted 2013-02-26; First posted 2013-04-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Spinal Cord Injury.
Keywords: Spinal Cord Injury stem cell
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell [ MNCs ] (Other): transplantation of autologous stem cell [MNCs ]
  Interventions: Biological: Transplantation of Autologous stem cell [MNCs] .

INTERVENTIONS:
Biological: Transplantation of Autologous stem cell [MNCs] . — Intra thecal transplantation of Autologous stem cell [MNCs],100millions per dose in 3 divided doses at interval of 10 days.
  Other Names: Autologous stem cell[MNCs] .

SUMMARY:
This Study is a single arm,Phase I/II , single centre trial to check active comparing the safety and efficacy of Bone marrow derived autologous cell(100 million per dose) trial to be conducted for 36 months.

DETAILED DESCRIPTION:
A spinal cord injury (SCI) refers to any injury to the spinal cord that is caused by trauma instead of disease.[1] Depending on where the spinal cord and nerve roots are damaged, the symptoms can vary widely, from pain to paralysis to incontinence.[2][3] Spinal cord injuries are described at various levels of "incomplete", which can vary from having no effect on the patient to a "complete" injury which means a total loss of function.Injuries at any level can cause:Increased muscle tone (spasticity),Loss of normal bowel and bladder control (may include constipation, incontinence, bladder spasms),Numbness,Sensory changes Pain,Weakness, paralysis. This Study is a single arm,Phase I/II , single centre trial to check active comparing the safety and efficacy of Bone marrow derived autologous cell(100 million per dose) trial to be conducted for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from Spinal cord injury.
* willingness to undergo bone marrow derived autologous cell therapy.
* patient those provide fully Informed consent form for the study.
* Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.
* traumatic Injury of spinal cord with complete or partial damage by MRI and Spinal cord injury level should be below C4

Exclusion Criteria:

* Patient with pre- existing or current systemic disease such as Lung, liver,(exception:history of uncomplicated hepatitis A)gastrointestinal,cardiac , immunodeficiency(HIV)
* History of life threatening allergic or immune - mediated reaction.
* haemodynamically unstable patients.
* patient suffer from peripheral muscular dystrophy.
* lactating and pregnant woman
* alcohol drug abuse /dependence
* positive test result for hepatitis A and Hepatitis B OR C
* Major-traumatic brain injury and patient with psychiatric illness .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in overall sensory for motor control using Frankel score. | 6 month

SECONDARY OUTCOMES:
Improvement in pain sensation and Significant changes in Muscle Tones from base line | 6 month
-Improvement in sensory and motor dysfunction using ASIA( American spinal cord injury association ) Scale | 6 month
Significant changes in Muscle Tones and Improvement in pain sensation from base line | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India